CLINICAL TRIAL: NCT04555239
Title: Treatment of Subacute and Chronic Extremity Pain With Fascial Distortion Model (FDM) in the Emergency Department
Brief Title: FDM for Subacute and Chronic Extremity Pain in the ED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit sufficient numbers due to the pandemic
Sponsor: Carilion Clinic (Other)
Collaborators: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20-780
Record Dates: First submitted 2020-08-26; First posted 2020-09-18 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2021-04

CONDITIONS: Myofascial Pain; Chronic Pain; Extremities Disorders; Osteopathic Manipulation
MeSH Terms: conditions — Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care, Upper Extremity Pain (Active Comparator): Patients will receive standard emergency department care as determined by their treating physician for their extremity pain.
  Interventions: Other: Standard Care
- Standard of Care, Lower Extremity Pain (Active Comparator): Patients will receive standard emergency department care as determined by their treating physician for their extremity pain.
  Interventions: Other: Standard Care
- FDM, Upper Extremity Pain (Experimental): Patients will receive the FDM intervention for their extremity pain. They may also receive standard emergency department care as determined by their treating physician for their extremity pain.
  Interventions: Procedure: Fascial Distortion Model (FDM); Other: Standard Care
- FDM, Lower Extremity Pain (Experimental): Patients will receive the FDM intervention for their extremity pain. They may also receive standard emergency department care as determined by their treating physician for their extremity pain.
  Interventions: Procedure: Fascial Distortion Model (FDM); Other: Standard Care

INTERVENTIONS:
Procedure: Fascial Distortion Model (FDM) — Only treatment of herniated trigger points, continuum distortions, and/or trigger bands will be performed.
  * Herniated trigger points are single areas of sharp pain within soft tissue.
  * Continuum distortions are single points of sharp pain overlying bony tissues.
  * Trigger bands are lines of pain overlying either soft or bony tissues.
  Treatment with FDM is performed using firm, direct pressure over the area of the patient's pain with the provider's thumb. This pressure is applied at a single point or area indicated by the patient for herniated trigger points and continuum distortions, and along the indicated line of pain for trigger bands.
  Arms: FDM, Lower Extremity Pain; FDM, Upper Extremity Pain
Other: Standard Care — The usual standard of care for extremity pain varies from provider to provider and varies from patient to patient depending upon their comorbidities but often includes some combination of the following:
  * X-rays, if suspicion for fracture exists
  * Venous duplex ultrasound, if suspicion for DVT/SVT exists
  * Computed tomography (CT) angiogram (CTA), if suspicion for arterial occlusion exists
  * C-reactive Protein (CRP)/erythrocyte sedimentation rate (ESR)/arthrocentesis is suspicion if suspicion for septic arthritis exists
  * Arthrocentesis if suspicion for gout exists
  * Splinting/casting/immobilization
  * NSAIDs, Tylenol, or opioids for pain control
  * Possibly trigger point injections
  * Possibly osteopathic manipulation
  * Recommendations to use RICE (rest, ice, compression, elevation) at home
  * Physical/occupational therapy referral
  * Orthopedic referral

SUMMARY:
STUDY PURPOSE: To identify whether a low-cost, minimally invasive, one-time manual medicine intervention (fascial distortion model, FDM) is effective for the management of subacute and chronic extremity pain in the emergency department (ED). Demonstration of benefit may have far-reaching implications including reduction of pain medication use in the ED, shortened ED visit times, and future use of this intervention in the outpatient setting for chronic pain management.

METHODS: We plan to conduct a randomized, unblinded clinical trial of FDM for the management of subacute and chronic extremity pain. 296 patients ages 18 and older seeking care in the ER for extremity pain that has been present for more than one week and less than three months will be recruited from four emergency departments within the Carilion Clinic hospital network over a 3-year time period. Patients are recruited into the study by treating clinicians in the ER and must describe their pain according to a pattern amenable to treatment with FDM: a. Single point of sharp pain overlying soft tissues correlating to a herniated trigger point; b. Single point of sharp pain overlying bone correlating to a continuum distortion; c. Line or band of pain overlying soft tissues or bone correlating to a trigger band.

POPULATION: Adult patients presenting to Carilion Franklin Memorial Hospital (CFMH), Carilion New River Valley Hospital (CNRVH), Carilion Roanoke Memorial Hospital (CRMH), and Carilion Stonewall Jackson Hospital (CSJH). Prisoners and patients with known serious psychiatric comorbidities are specifically excluded.

Specific Aims: The primary objective is to determine whether FDM yields significant improvement in function compared with standard care alone. The secondary objective is to determine whether FDM yields significant improvement in pain compared with standard care alone. Our exploratory objective is to determine whether FDM yields clinically significant improvements in pain and function that endure over time.

HYPOTHESIS: Patients treated with FDM will demonstrate statistically and clinically significant improvement in function and pain compared with those treated with standard care alone.

SIGNIFICANCE: This is the first clinical trial of FDM in the United States and the first in an ED.

DETAILED DESCRIPTION:
The application of FDM for the treatment of non-specific subacute and chronic extremity pain in the ED combined with standard care holds enormous promise. High-quality studies investigating whether single-episode FDM therapy in the ED is effective are needed. Our goal is to conduct a randomized, prospective clinical trial investigating the use of FDM plus standard ED pain management for non-specific subacute and chronic extremity compared with standard ED pain management.

The anticipated outcome of this study is statistically and clinically significant improvement in function and pain in those treated with FDM compared with those compared with standard emergency department care alone for their extremity pain. Demonstration of such results would provide stronger evidence base for manual manipulation, particularly in the emergency department setting. This is a low-cost intervention that can be learned easily by physicians and providers of a variety of backgrounds (advanced care practitioners, physical therapists, etc.) and can thus provide an excellent alternative for pain management as opposed to our traditional approaches to pain such as rest, ice, compression, and elevation (RICE), and medications such as NSAID (non-steroidal anti-inflammatory drugs) and acetaminophen. We all realize that part of the reason we are struggling with an opioid epidemic in our country is that our traditional approaches to pain management are not always enough and that patients subsequently become dependent upon stronger medications for pain control that unfortunately have addictive properties as side effects. If FDM proves to be a successful intervention for managing subacute and chronic pain in the emergency department with a single treatment, imagine its applicability on a wider scale in the outpatient setting for chronic pain management and how this could help us combat the current opioid crisis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 and older with arm or leg pain for which they are presenting to the emergency department.
2. Pain has been present for greater than one week and less than three months.
3. Pain is described in terms amenable to treatment by FDM:

   * Single point of sharp pain overlying soft tissues correlating to a herniated trigger point.
   * Single point of sharp pain overlying bone correlating to a continuum distortion.
   * Line or band of pain overlying soft tissues or bone correlating to a trigger band.
4. Patient is able to speak, read, and write fluently in the English language.
5. Patient is able to be reached by telephone for follow up.
6. Patient has access to text messaging services, email, and the internet.

Exclusion Criteria:

1. Inability to make informed consent (i.e. cognitive impairment or untreated psychiatric illness that would prohibit the ability to comprehend the risks and benefits of manipulative treatment vs. standard treatment).
2. Location of pain overlies major neurovascular structures (which would thus inhibit direct manipulation in that area).
3. Chronic systemic illness or medication treatment that would make patients prone to prolonged bruising or significant swelling after manipulation, including:

   * Active chemotherapy or radiation treatment.
   * Chronic steroid use.
   * Chronic wounds due to vascular disease or diabetes.
   * End stage renal disease on dialysis (risk of calciphylaxis).
   * Immunocompromised status.
   * Lymphedema.
   * Venous stasis insufficiency.
4. Connective tissue diseases, such as Marfan's or Ehlers-Danlos.
5. Dermatologic conditions:

   * Fragile skin that would be prone to tears with manipulation.
   * Skin lesions including open wounds or rashes overlying area of pain.
6. Neurologic conditions:

   * Peripheral neuropathy limiting sensation in the area of pain.
   * Demyelinating disease involving the extremity where the pain is located.
7. Orthopedic conditions:

   * Joint replacement underlying location of pain.
   * Prior orthopedic surgery to the area of pain.
   * Fracture, known or suspected, underlying site of pain.
8. Vascular conditions:

   * Superficial venous thrombosis (SVT), thrombophlebitis, or deep venous thrombosis (DVT) or suspicion for these underlying site of pain.
   * Current treatment with anticoagulants other than aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Statistically Significant Functional Improvement | 6 months
  To determine whether a single FDM treatment provided in the ED yields significant improvement in function for patients with subacute and chronic extremity pain, and whether this effect endures over time.

SECONDARY OUTCOMES:
Statistically Significant Pain Improvement | 6 months
  To determine whether a single FDM treatment provided in the emergency department yields significant improvement in pain for patients with subacute and chronic extremity pain, and whether this effect endures over time.

OTHER OUTCOMES:
Clinically Significant Functional Improvement | 6 months
  Whether FDM yields clinically significant improvements in function that last over time.
  - Clinical significance is defined as a change of at least 11 points on the Disabilities of the Arm, Shoulder, and Hand (DASH) Score from baseline or change of at least 9 points on the Lower Extremity Functional Scale (LEFS) Score from baseline.
Clinically Significant Pain Improvement | 6 months
  Whether FDM yields clinically significant improvements in pain pre-intervention that last over time. [Clinical significance is defined as 13 mm or greater improvement in visual analogue scale (VAS) score.]

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Bernier, D.O., Principal Investigator — Carilion Clinic
Locations (4):
- United States (4):
  - Carilion New River Valley Medical Center, Christiansburg, Virginia
  - Carilion Stonewall Jackson Hospital, Lexington, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Carilion Franklin Memorial Hospital, Rocky Mount, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capistrant, Todd A., and Steve LeBeau. Why Does It Hurt?: the Fascial Distortion Model: a New Paradigm for Pain Relief and Restored Movement. Beaver's Pond Press, 2014.
- [Background] Fink M, Schiller J, Buhck H. [Efficacy of a manual treatment method according to the fascial distortion model in the management of contracted ("frozen") shoulder]. Z Orthop Unfall. 2012 Sep;150(4):420-7. doi: 10.1055/s-0032-1314996. Epub 2012 Aug 23. German. PMID 22918828
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Schulze C, Finze S, Bader R, Lison A. Treatment of medial tibial stress syndrome according to the fascial distortion model: a prospective case control study. ScientificWorldJournal. 2014;2014:790626. doi: 10.1155/2014/790626. Epub 2014 Oct 14. PMID 25379543
- [Background] Boucher JD, Figueroa J. Restoration of Full Shoulder Range of Motion After Application of the Fascial Distortion Model. J Am Osteopath Assoc. 2018 May 1;118(5):341-344. doi: 10.7556/jaoa.2018.044. PMID 29507951
- [Background] Richter D, Karst M, Buhck H, Fink MG. Efficacy of Fascial Distortion Model Treatment for Acute, Nonspecific Low-Back Pain in Primary Care: A Prospective Controlled Trial. Altern Ther Health Med. 2017 Sep;23(5):AT5522. Epub 2017 Jun 23. PMID 28646809
- [Background] Hsu JR, Mir H, Wally MK, Seymour RB; Orthopaedic Trauma Association Musculoskeletal Pain Task Force. Clinical Practice Guidelines for Pain Management in Acute Musculoskeletal Injury. J Orthop Trauma. 2019 May;33(5):e158-e182. doi: 10.1097/BOT.0000000000001430. PMID 30681429
- [Background] Abdolrazaghnejad A, Banaie M, Tavakoli N, Safdari M, Rajabpour-Sanati A. Pain Management in the Emergency Department: a Review Article on Options and Methods. Adv J Emerg Med. 2018 Jun 24;2(4):e45. doi: 10.22114/AJEM.v0i0.93. eCollection 2018 Fall. PMID 31172108
- [Background] National Center for Health Statistics. "National Hospital Ambulatory Medical Care Survey: 2016 Emergency Department Summary Tables." CDC.gov, 2016, www.cdc.gov/nchs/data/nhamcs/web_tables/2016_ed_web_tables.pdf.
- [Background] Thalhamer C. A fundamental critique of the fascial distortion model and its application in clinical practice. J Bodyw Mov Ther. 2018 Jan;22(1):112-117. doi: 10.1016/j.jbmt.2017.07.009. Epub 2017 Jul 25. PMID 29332733
- [Background] Eisenhart AW, Gaeta TJ, Yens DP. Osteopathic manipulative treatment in the emergency department for patients with acute ankle injuries. J Am Osteopath Assoc. 2003 Sep;103(9):417-21. PMID 14527076
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Gould D, Kelly D, Goldstone L, Gammon J. Examining the validity of pressure ulcer risk assessment scales: developing and using illustrated patient simulations to collect the data. J Clin Nurs. 2001 Sep;10(5):697-706. doi: 10.1046/j.1365-2702.2001.00525.x. PMID 11822520
- [Background] "Writing a Protocol." Writing a Protocol | CHOP Institutional Review Board, 2019, irb.research.chop.edu/writing-protocol.